CLINICAL TRIAL: NCT04789226
Title: Psychological Impact of Covid-19 Assiut University Hospital Experience
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Yassin Ibrahim, Principal investigator, Assiut University
Other Study IDs: Psychology and covid 19
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Psychological Impact of Covid-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psychological impact of covid-19 in assiut university hospital

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is a new communicable disease caused by the new strains of severe acute respiratory syndrome coronavirus, SARS-CoV-2 . The first outbreak reported was in December2019, in Wuhan, China, as pneumonia of unknown etiology linked to a seafood market exposure COVID-19 affects different people in different ways. Most infected people will develop mild to moderate illness and recover without hospitalization.

The evolution of the novel Corona Virus Disease (COVID-19) and its expeditious dissemination have led the World Health Organization (WHO) to declare it a pandemic on 11 March 2020 . As of 16 May 2020, there have been 4,425,485 confirmed COVID-19 cases and 302,059 related deaths worldwide and Egypt has been among the most affected countries in the Eastern Mediterranean region with 11,228 confirmed cases and 592 deaths .

As a consequence, many countries, including Egypt, have set a state of lockdown to hinder the spread of infection among people resulting in a global atmosphere of depression and anxiety associated with social isolation, fears of getting infected, breaks in the supply chains, financial distress, disrupted travel plans, and future uncertainty . Several epidemiological studies from China detected a high prevalence of psychological disturbances among the public during the COVID-19 pandemic. For example, a large online survey of 56,679 individuals from 34 provinces in China reported numerous psychological conditions during the COVID-19 pandemic: depression (27.9%), anxiety (31.6%), stress (24.4%), and insomnia (29.2%) . Also, a study conducted on 4872 Chinese people from 31 provinces showed a high prevalence of depression (48.3%) and anxiety (22.6%) related to the COVID-19 pandemic . A similar study revealed depression (20.1%), anxiety (35.1%), and poor sleeping (18.2%) among 7236 Chinese people . Another study conducted on 7143 college students in China detected anxiety among 25% of them .

In low- and middle-income countries, such as Egypt, where infection control precautions, surveillance programs, laboratory capacity, and public health resources are limited , the response to the COVID-19 pandemic is challenging and, as a result, the psychological impacts of the pandemic on the public can be even worse. Thus, we conducted this study to evaluate several forms of psychological disturbances .

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years old
* diagnosed as covid-19 by positive PCR
* comes to Assiut University Hospital
* both sex males and females

Exclusion Criteria:

* age less than 18 years old
* past history of psychatric disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients more than 18 years old and less than 90 years old diagnosed as covid-19 by positive PCR
Sampling Method: Non-Probability Sample
Enrollment: 239 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Symptom Checklist 90 "SCL 90" | One year
  it is a 90 item questionnaire used to assess psychological problems .
post traumatic stress disorder "PTSD" | One year
  PCL-5 is a 20 item self report measure that assesses the 20 DSM-5 symptoms of PTSD .
Pittsburgh Sleep Quality Index "PSQI" | One year
  evaluating sleep quality in older adults , the pittsburgh sleep quality index can be used to detect sleep disturbance or deficits .
The 36- items Short Form"SF 36" | one year
  consists of eight scaled scores , which are the weighted sums of the questions in their section " evaluating individual patients health status " .